CLINICAL TRIAL: NCT04375683
Title: A Study of Efficacy and Safety of Flumatinib Combined With Chemotherapy in the Treatment of Ph Positive Acute Lymphoblastic Leukemia Based on Minimal Residual Disease Monitoring
Brief Title: Study of Efficacy and Safety of Flumatinib Combined With Chemotherapy in Ph Positive ALL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Ge Zheng, Principal Investigator, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDYYGZ202003
Record Dates: First submitted 2020-04-26; First posted 2020-05-05 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Acute Lymphocytic Leukemia, Adult B-Cell; BCR-ABL1 Fusion Protein Expression
Keywords: Flumatinib; minimal residual disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — flumatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ph-positive ALLs (Experimental): Subjects aged 60 years or older are received flumatinib and dose-adjusted VDCP or prednisone regimen. Subjects younger than 60 years are received flumatinib and hyper-CVAD regimen
  Interventions: Drug: Flumatinib

INTERVENTIONS:
Drug: Flumatinib — Flumatinib 600mg per day, taken on empty stomach

SUMMARY:
Philadelphia chromosome (BCR-ABL1, Ph) is the most common genetic abnormality in acute lymphoblastic leukemia (ALL) and an independent prognostic risk factor. With the increase of age, the incidence of patients over 60 years old can reach 50%, whose 5-year overall survival rate was less than 20%.

With the application of tyrosine kinase inhibitor (TKI), the prognosis of Ph positive ALL patients is greatly improved. At present, TKI combined with chemotherapy has become the first-line treatment recommended in the guideline of Ph positive ALL patients.

However, with the use of imatinib, more and more patients develop drug resistant to imatinib. In addition, the clinical data showed that the MRD negative rate in patients treated with imatinib combined with hyper CVAD was only 22% three months later, which was far lower than 31% of the second generation TKI and 52% of the third generation TKI.

Second generation TKI dasatinib and nilotinib can overcome most imatinib resistant kinase region mutations. However, patients with severe hemocytopenia, infection or other complications are often unable to tolerate the standard chemotherapy. In addition, due to the high cost, some patients can't afford the long-term use.

Flumatinib is the first approved second generation TKI in China and a derivative of imatinib. Compared with imatinib, it introduced trifluoromethyl, substituted pyridine ring for benzene ring, and kept the direction of amide bond, which made the inhibitory effect of flumatinib on common kinase mutations significantly better than that of imatinib. In addition, compared with the second-generation TKI recommended in the first line of current guidelines, the incidence of quality of life related adverse reactions of flumatinib is lower, and no specific adverse reactions of the second-generation TKI have been reported.

We plan to enroll 28 patients with Ph positive ALL. All patients are diagnosed by morphology, immunology, cytogenetics and molecular biology (MICM). According to subjects' age, we will divide them into two groups. Subjects aged 60 years or older are received flumatinib and dose-adjusted VDCP or prednisone regimen. Subjects younger than 60 years are received flumatinib and hyper-CVAD regimen. MRD are examined on the 8th, 15th and 29th day after chemotherapy. Then, MRD will be monitored in the third, 6th, 9th, 12th, 15th, 18th, 21th and 24th months after chemotherapy to evaluate the effect.

DETAILED DESCRIPTION:
Flumatinib + hyper-CVAD (younger than 60):

Induction therapy: Flumatinib 600mg per day, on an empty stomach; For cycles 1, 3, 5, and 7: cyclophosphamide (CTX) 300 mg/m² is given intravenously over 3 h every 12 h for six doses on days 1-3; a continuous daily infusion of sodium mercaptoethanesulfonate (Mesna) at 600 mg/m² per day for 24h starting 1h before CTX and completed approximately 12h after the final CTX dose; doxorubicin 50 mg/m² is given intravenously over 24 h on day 4; vincristine (VCR) 1.4 mg/m² (Maximum daily dose 2 mg) is intravenously on days 4 and 11; dexamethasone (Dex) 40 mg is given intravenously or orally on days 1-4 and days 11-14. For cycles 2, 4, 6, and 8: methotrexate (MTX) is given intravenously at 200 mg/m² over 2 h, followed by 800 mg/m² over 22 h on day 1; cytarabine (Ara-C) 3 g/m² is given intravenously over 3 h every 12 h for four doses on days 2-3; citrovorum 50 mg is given intravenously, followed by 15 mg every 6 h for eight doses beginning 12 h after MTX completion. Prophylactic intrathecal therapy will be given after complete remission.

Maintenance therapy (given for 2 years): intravenous VCR 1.4 mg/m² on day 1 (Maximum daily dose 2 mg), every three months; oral dexamethasone 8mg/m² on days 1-7, every three months; oral 6-MP 60mg/m² on days 1-7, every month; oral MTX 20mg/m² on day 8, every month; and daily flumatinib at 600 mg. Months 6 and 13 of maintenance were intensification courses of hyper-CVAD and flumatinib.

Flumatinib + dose-adjusted VDCP (fit group, 60 years or older):

Induction therapy: flumatinib 600mg per day, on an empty stomach; vincristine (VCR) 1.4mg/m2/d (maximum daily dose 2mg) is given intravenously on day 1, 8, 15, 22; daunorubicin (DNR) 30mg/m2/d is given intravenously on day 1, 8, 15, 22 (if blasts of day 15 lower than 20%, DNR is not needed on day 15 and 22); cyclophosphamide (CTX) 400mg/m2/d is given intravenously on day 1,8,15 and 22; Prednisone 60mg/m2/d is given orally every other day for day 1-22. Prophylactic intrathecal therapy will be given after complete remission.

Consolidation therapy: flumatinib 600mg per day; daunorubicin (DNR) 40mg/m2 is given intravenously on day 1; cytarabine (Ara-C) 60mg/m2 is given intravenously on day 1-5; L-Asparaginasum (L-Asp) 500U/kg is given intravenously on day 6-10. If complete remission (CR) on day 28, a consolidation chemotherapy will be given on day 35; if not, we will give it as salvage therapy; And if CR is achieved after salvage therapy, another consolidation chemotherapy will be given.

Maintenance therapy (given for 2 years): intravenous VCR 1.4 mg/m² on day 1 (Maximum daily dose 2 mg), every three months; oral dexamethasone 8mg/m² on days 1-7, every three months; oral 6-MP 60mg/m² on days 1-7, every month; oral MTX 20mg/m² on day 8, every month; and daily flumatinib at 600 mg.

Flumatinib + Prednisone (unfit group, 60 years or older):

Prephase: Prednisone 60 mg/m2/d po, Day -7 to day -1. Induction therapy: flumatinib 600mg per day, on an empty stomach; Prednisone 60 mg/m2 per day day 1-24 and then tapered and stopped at day 32.

Maintenance therapy (given for 2 years): flumatinib 600mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Ph positive ALL
* Signing informed consent voluntarily

Exclusion Criteria:

* Severe mental disorder
* Uncontrolled heart disease
* Be allergic to flumatinib or other research drugs
* More than 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | day 28
  blasts in bone marrow are less than 5%
minimal residual disease | Change from MRD at 2 years
  MRD is measured by flow cytometry and qPCR

SECONDARY OUTCOMES:
side effects | 6 months
  Number of participants with bone marrow suppression, nausea and vomiting, diarrhea, infection, and non-hematologic toxicity such as heart, liver, kidney and nervous system damage

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Ge, PhD. MD., Study Chair — Zhongda Hospital
Locations (1):
- Department of Hematology, Zhongda Hospital Southeast University, Institute of Hematology Southeast University, Nanjing, Jiangsu, China